CLINICAL TRIAL: NCT03647631
Title: Sentinel Lymph Node Biopsy in Porocarcinoma: A Case Reports
Brief Title: Sentinel Lymph Node Biopsy in Porocarcinoma
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Other Study IDs: Chirurgia1
Record Dates: First submitted 2018-08-17; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Porocarcinoma; Sentinel Lymph Node
MeSH Terms: conditions — Eccrine Porocarcinoma | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients affected to porocarcinoma
  Interventions: Procedure: sentinel lymph node biopsy
- patients affected to porocarcinoma in our centre
  Interventions: Procedure: sentinel lymph node biopsy

INTERVENTIONS:
Procedure: sentinel lymph node biopsy — Authors discuss a possible usefulness of SNLB for staging and diagnosis in porocarcinoma.

SUMMARY:
Eccrine porocarcinoma (EPC) is a slow-growing carcinoma arising from the eccrine sweat glands. Based on its clinical presentation it can be confused with malignant and benign skin lesions, both. Histological examination is essential to formulate a correct diagnosis. Surgical excision with clear margins is the standard therapeutic approach while the role of sentinel lymph node biopsy (SNLB) remains controversial.

The Authors report two cases of EPC of the lower limbs occurred in two women. Patients were treated by wide surgical excision of the lesion and SNLB.

DETAILED DESCRIPTION:
INTRODUCTION Eccrine porocarcinoma (EPC), first described by Pinkus and Mehregan in 1963, is a rare form of skin cancer. Its presentations very often mimics a cutaneous lesion similar to other forms of benign and malignant cutaneous neoplasms. Accurate diagnosis, optimal treatment and prognosis of EPC are still challenging due to scant literature reports. Eccrine carcinomas may have an elevate presence of regional lymph node metastasis, thus some authors have advocated SLNB for all or some patients, but its utility for staging purposes remains unknown.

We report two cases of EPC in which the sentinel lymph node biopsy (SLNB) was performed.

CASE PRESENTATION Case 1 During August 2017, a 64 years woman was seen at our department after a previous cutaneous lesion excision with an histological diagnosis of porocarcinoma of the left thigh. The histological examination revealed a poroid neoplasm extending into the deep dermis to the level of the dermal-subcutaneous junction with a thickness of 5.4mm, 10-12 mitoses per 10 high-power field, absence of lymphovascular invasion and free margins with a clearing distance of 1.5 mm. Hematoxilyn-eosin staining and Immunohistochemical (IHC) analysis showed positive staining for carcinoembryonic antigen (CEA), cytokeratin (CK) 5,7 and epithelial membrane antigen (EMA).

She had a past medical history of appendicitis in childhood, anxious-depressive syndrome, osteoporosis, hiatal hernia, obesity and smoked about 20 cigarettes a day. New York Heart Association (NYHA) score was 1 and American Society of Anesthesiologists (ASA) score was 1. The patient had no anorexia and weight loss and the examination did not reveal any inguinal lymphadenopathy. Laboratory tests, including blood count, biochemical investigations and serological viral markers were normal. The electrocardiogram showed sinus rhythm and the chest radiograph showed no signs of pleural or parenchymal lesions. After multidisciplinary discussion and based on the sub-optimal clearing margin we performed a re-excision of the previous wound to ensure wider safety margins of at least 20 mm similarly to surgical strategy for other skin tumors and in particular melanoma. At that time it was also decided to perform a SLNB; preoperative lymph-node scintigraphy showed the presence of two sentinel lymph nodes in the left groin that were excised during SLNB.

Case 2 During August 2017, a 65year-old female was admitted to our department with histological finding of EPC of the right leg. One month before, she underwent surgical excision of a cutaneous lesion of the right leg. This lesion appeared brownish, exophytic, with ulcerated surface, more suggestive for a squamous cell carcinoma than an ulcerated nodular basal cell carcinoma. The histological examination revealed a poroid neoplasm extending into the reticular dermis with a thickness of 5 mm, 10 mitoses per 10 high-power field, absence of lymphovascular invasion and free margins with a clearing distance of 2 mm.

She had a past medical history of hysterectomy and bilateral salpingo-oophorectomy for uterine fibromatosis, kidney transplantation for severe chronic renal failure, high blood pressure, aneurysmal dilatation of the right common carotid artery, hypercholesterolemia, hyperparathyroidism and previous inferior myocardial infarction. Laboratory tests, including blood count, biochemical investigations and serum viral markers were normal. After multidisciplinary discussion and based on the sub-optimal clearing margin we performed a re-excision of the previous wound to ensure wider safety margins of at least 20 mm. It was also decided to perform a SLNB; the pre-operative lymph node scintigraphy showed the presence of two sentinel lymph nodes in the right inguinal site. The patient underwent enlargement of the surgical excision until 20 mm of free margin from the previous excision and SLNB of the two lymph nodes identified preoperatively.

DISCUSSION EPC is a rare neoplasm arising from the intra-epidermal ductal portion of the eccrine sweat gland and represents approximately 0.005 % of all cases of malignant epithelial neoplasms.

Elderly patients are the most affected, with a peak incidence between the 6th and7th decade of life. Although it does not seem to have a predilection for sex or race, some studies indicate a slight prevalence in women. The exact etiology of EPC is unclear. Some authors suggested a possible association with radiation exposure and immunosuppression although an excessive sun exposure does not seem to be a significant risk factor. EPC may arise de novo or can develop from a pre-existing benign lesion; some clinical signs, such as spontaneous bleeding, sudden growth and ulceration in a longstanding stable lesion must lead to the suspicion of malignant degeneration. Clinically EPC can be presented as an erythematous or violaceous nodule, papule or plaque with an infiltrative or erosive pattern. EPC usually arises on the lower extremities (44%), followed by the trunk (24%), head & neck (23%), upper extremities (11%), and rarely involves other areas. Microscopically, EPC is characterized by a cluster of anaplastic cells with nuclear hyperchromasia and important mitotic activity, extending from the epidermis to the dermis, surrounded by ductal lumen. Robinson et al. reported specific histopathologic features of EPC which may be predictive of a less favorable outcome. Thickness is the main prognostic factors for EPC. Tumors greater than 7 mm in thickness, an infiltrating front of tumor cells, the presence of lymphovascular invasion, and greater than 14 mitoses per high-power field were noted to be associated with a poorer prognosis.

The differential diagnosis includes basal and squamous cell carcinoma, adenocarcinoma, amelanotic melanoma, Bowen's disease, Paget's disease and also benign lesions like fibroma and pyogenic granuloma. Some immunohistochemical markers as carcinoembryonic antigen (CEA), EMA, and p53 protein may play a role in the diagnosis of EPC.

Therapeutic options for the treatment of EPC include electrofulguration, electrocautery, surgical excision, radiation and amputation. Surgical excision with histologically clear margins is generally considered the treatment of choice with cure rates as high as 70-80 %, although a recurrence rate of up to 20% has been reported. This elevate incidence of local recurrence may be due to a not optimal free margin at surgical excision. Lymph node metastases are present at diagnosis in 20% of cases and the incidence of visceral metastases is reported to be 10%. The tumor tends to spread tangentially in the lower third of the epidermis, then after infiltrates the dermis, subcuticular fat and lymphatic system. The role of sentinel lymph node biopsy remains controversial.

ELIGIBILITY:
patients affected to moderate and high risk porocarcinoma, in according to hystophatological findings, submitted to SNLB.

Inclusion criteria:

1. Thickness greater than or equal to 5mm
2. mitoses per 10 high-power field greater than or equal to 7
3. Immunohistochemical (IHC) analysis positive for :carcinoembryonic antigen (CEA), cytokeratin (CK) 5,7 and epithelial membrane antigen (EMA).
4. Informed consent obtained for the SNLB procedure.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: two cases of EPC in which the sentinel lymph node biopsy (SLNB) was performed.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Role of SNLB in porocarcinoma in two patients evaluating the percentage of positive lymph nodes removed. | Patients were treated by wide surgical excision of the lesion and SNLB. 6 months follow-up was the time frame of the study.
  The investigators evaluated the role of SNLB in patients affected to moderate and high risk porocarcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Palombo, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No